CLINICAL TRIAL: NCT01717560
Title: Hepatitis C Treatment in Underserved Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Brian Edlin (Other)
Collaborators: Weill Medical College of Cornell University (Other); State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor-Investigator, Brian Edlin, Associate Professor of Medicine and Public Health, Weill Medical College of Cornell University
Organization: Weill Medical College of Cornell University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0308006281
Record Dates: First submitted 2008-04-29; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Hepatitis C; Illicit Drug Use
Keywords: chronic hepatitis C; illicit drug use; Substance-Related Disorders; multidisciplinary care; integrated care; mental health care; intensive case management
MeSH Terms: conditions — Hepatitis C, Chronic; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Collaborative multidisciplinary integrated care (Experimental): Collaborative, multidisciplinary, integrated care for hepatitis C
  Interventions: Other: Collaborative, multidisciplinary, integrated care

INTERVENTIONS:
Other: Collaborative, multidisciplinary, integrated care — Collaborative, multidisciplinary, integrated care for hepatitis C
  multidisciplinary model that combines expert care in five domains: (a) antiviral pharmacotherapy for HCV infection; (b) substance abuse treatment; (c) psychiatric evaluation and treatment; (d) primary medical care; and (e) intensive, client-centered, case management.

SUMMARY:
The purpose of this study is to examine the feasibility, safety, and effectiveness of treating persons who are actively using illicit drugs for hepatitis C using a collaborative, multidisciplinary, integrated care model. We hypothesize that by maximizing facilitators and minimizing barriers to treatment we can enable drug users to receive effective treatment for hepatitis C.

DETAILED DESCRIPTION:
This study examines the feasibility of integrated treatment for hepatitis C in active IDUs using a client-centered, multidisciplinary model that combines expert care in five domains: (a) antiviral pharmacotherapy for HCV infection; (b) substance abuse treatment; (c) psychiatric evaluation and treatment; (d) primary medical care; and (e) intensive, client-centered, case management. The Weill Cornell Medical College Center for the Study of Hepatitis C collaborates with community-based organizations providing services to injection drug users to provide multidisciplinary, integrated care using a model that combines the resources of culturally appropriate community-based agencies with those of a state-of-the-art tertiary care center.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Used heroin, cocaine, or injected other drugs for at least 1 year
* Have used heroin, cocaine and/or methamphetamine within the last 30 days
* Test positive for HCV antibody
* Are interested in being evaluated for HCV treatment

Exclusion Criteria:

* Persons who are obviously intoxicated, incoherent or otherwise unable to give informed consent are excluded from participation. Such persons may participate in the study if they return at a later date and are capable of providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-02; Primary Completion 2012-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Sustained virologic response, defined as an undetectable serum HCV RNA level 24 weeks after completion of antiviral therapy. | 24 weeks after completion of antiviral treatment
  SVR is measured 24 weeks after completion of antiviral treatment

SECONDARY OUTCOMES:
completion of medical and psychiatric evaluation for antiviral therapy | Patients are expected to complete medical and psychiatric evaluation within 3-6 months but it may take longer in some cases.
initiation of antiviral therapy | Patients are expected to initiate antiviral therapy (or decide not to) within 3-6 months but it may take longer in some cases.
adherence to antiviral therapy | Weekly up to 48 weeks
  Adherence is measured weekly during the duration of prescribed antiviral therapy. (Antiviral therapy is prescribed for up to 48 weeks, depending on the patient's characteristics, the regimen, and the response to therapy.)
completion of antiviral therapy | Completion is recorded at the time prescribed antiviral therapy is discontinued, whether that happens when the prescribed duration of therapy is complete or before. (Antiviral therapy is prescribed for up to 48 weeks, depending on the patient.)
levels of alcohol and illicit drug use | Weekly up to 96 weeks
  Measured weekly during antiviral therapy and monthly before and after therapy for the duration of follow-up
entry into treatment for substance use | Monthly up to 24 months
  Measured monthly from study enrollment through 24 weeks subsequent to completing prescribed course of antiviral therapy
entry into treatment for another unaddressed medical or psychiatric condition | Monthly up to 24 months
  Measured monthly from study enrollment through 24 weeks subsequent to completing prescribed course of antiviral therapy
neuropsychiatric side effects, including depression and hostility/irritability | Monthly up to 72 weeks
  Measured monthly during prescribed course of antiviral therapy and for 24 weeks thereafter
treatment-limiting systemic, hematologic, or other side effects | Weekly up to 72 weeks
  Measured weekly during prescribed course of antiviral therapy and then monthly or quarterly thereafter (TSH, for example, is measured every 3 months during and after treatment)
other adverse events or adverse effects | Monthly up to 72 weeks
  Measured monthly during prescribed course of antiviral therapy or as patients bring adverse events or effects to attention of physicians or study staff
reinfection | Quarterly up to 10 years
  Patients are monitored at 3-month intervals for reinfection. This will continue as long as possible after completion of antiviral therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Brian R. Edlin, MD, Principal Investigator — Weill Medical College, Cornell University
Locations (1):
- Center for the Study of Hepatitis C, Weill Medical College, Cornell University, New York, New York, United States